CLINICAL TRIAL: NCT06345885
Title: Immunogenicity and Safety of One Dose of Cecolin and One Dose of Gardasil
Brief Title: Immunogenicity and Safety of One Dose of HPV Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROPMHP002
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Human Papillomavirus Vaccines
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Bivalent HPV Vaccine (Cecolin)
  Interventions: Biological: HPV vaccine
- Group B (Active Comparator): Quadrivalent HPV vaccine (Gardasil)
  Interventions: Biological: HPV vaccine

INTERVENTIONS:
Biological: HPV vaccine — Participants in the group A will be administrated with bivalent HPV vaccine Cecolin. The immunization schedule is 0, 6 months; Participants in the group B will be administrated with quadrivalent HPV vaccine Gardssil. The immunization schedule is 0, 2, 6 months

SUMMARY:
This study will assess the immunogenicity and safety of one dose of Cecolin and one dose of Gardasil

ELIGIBILITY:
Inclusion Criteria:

* Female, aged between 9 and 14 years (including 9 and 14 years) on the day of enrollment
* Judged as healthy and eligible for vaccination by the investigators through a self- reported medical history and some physical examinations
* Subjects and legal guardians are informed and agree, and sign the Informed Consent Form
* Female urine pregnancy test is negative

Exclusion Criteria:

* Axillary temperature>37.2 ℃
* Other investigational or unregistered products (drugs or vaccines) that have been used or planned to be used during the study period within 30 days prior to receiving the research vaccine
* Systemic use of immunosuppressants or other immunomodulatory drugs or corticosteroids for a long period of time (lasting for more than 14 days) within 6 months prior to receiving the research vaccine, but local use is allowed (such as ointments, eye drops, inhalers, or nasal sprays)
* Within 3 months prior to vaccination, immunoglobulin and/or blood preparations were used or planned to be used during the study period, but emergency use of tetanus immunoglobulin and rabies immunoglobulin is allowed after exposure
* Received inactivated vaccines within 14 days prior to enrollment in the study, or received live vaccines within 21 days prior to enrollment in the study
* Fever (axillary temperature ≥ 38.0 ℃) within 3 days prior to vaccination, or any acute illness requiring systemic antibiotics or antiviral treatment within the past 5 days
* Previously received HPV vaccine
* Immunodeficiency diseases, chronic medical histories that require treatment for important organs such as primary diseases, cancer (or precancerous lesions), immune diseases (including systemic lupus erythematosus, rheumatoid arthritis, any condition leading to splenectomy or splenectomy, and other immune diseases that researchers believe may have an impact on immune response)
* Have a history of allergies, including serious adverse reactions from previous vaccination, such as allergies, urticaria, breathing difficulties, angiogenic edema, or abdominal pain
* Asthma, with unstable conditions in the past two years requiring emergency treatment, hospitalization, oral or intravenous corticosteroids
* Complicated with serious medical diseases, such as hypertension, heart disease, diabetes, hyperthyroidism, etc
* Abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or coagulation disorders diagnosed by doctors
* Epilepsy, excluding febrile epilepsy under 2 years old and simple epilepsy that did not require treatment in the past 3 years
* Due to the inability to comply with research requirements due to psychological conditions, having a past or present mental illness that has not been well controlled within the past two years, requiring medication for mental illness, and having suicidal tendencies in the past five years
* According to the researcher's judgment, due to various medical, psychological, social, occupational factors or other conditions, it is contrary to the research plan or affects the recipient and guardian to sign informed consent

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Anti-HPV seropositivity | At 1 month after first dose
  Seropositivity to HPV16 and HPV18 types of the neutralizing antibody in subjects will be assessed.

SECONDARY OUTCOMES:
Anti-HPV Seropositivity | At 2 months after first dose
  Seropositivity to HPV16 and HPV18 types of the neutralizing antibody in subjects will be assessed.
HPV Antibody Titers | At 1 and 2 months after first dose
  Geometric mean titers (GMT) of HPV16 and HPV18 types at 1 and 2 months after the first dose of vaccine administration in the subjects will be assessed.
Local and Systemic Reactions/Event | 7 and 30 days after each dose of vaccination; 0-7 months
  Soliciting local reactions/events; Soliciting systemic reactions/events; Non solicited adverse events; Serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Center for Disease Control and Prevention, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263